CLINICAL TRIAL: NCT00724282
Title: Double-blind Placebo-controlled Study of the Effects of Eszopiclone on Glucose Tolerance, Insulin Secretion, and Insulin Action in Adults With Chronic Insomnia
Brief Title: Treatment of Insomnia and Glucose Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15632; ESRC-124
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Sleep; Insomnia; Insulin Resistance
Keywords: sleep; eszopiclone; insulin secretion; insulin action; glucose tolerance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Insulin Resistance | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eszopiclone or Placebo (Other): Subjects receive either eszopiclone or placebo for 9 days, followed by 3 week washout, then crossover to opposite treatment. Treatment is double-blinded.
  Interventions: Drug: Eszopiclone; Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone 3 mg by mouth daily at bedtime for 9 days
  Other Names: Lunesta
Drug: Placebo — Placebo by mouth daily at bedtime for 9 days

SUMMARY:
Available data suggest that obtaining adequate sleep is associated with a better ability of the body to use carbohydrates as a source of energy and a lower risk of developing diabetes. The sleeping pill, Eszopiclone (Lunesta), has been approved by the Food and Drug Administration for the treatment of people who complain of trouble falling or staying asleep. This study will examine the hypothesis that the use of Eszopiclone (Lunesta) to improve the sleep of people with insomnia may also improve the use of sugar in their body.

DETAILED DESCRIPTION:
Study participants will complete a set of oral and intravenous glucose (sugar) tolerance tests, which will be performed on two separate occasions in random order: once after a week of treatment with Eszopiclone (Lunesta) and once again after a week of receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* age between 35 and 64
* must have long-standing trouble falling or staying asleep
* BMI between 22 and 34 kg/m2

Exclusion Criteria:

* sleep apnea or other sleep disorder other than insomnia
* diagnosis of diabetes requiring treatment with pills or insulin
* smoking
* night or shift work
* presence of a medical condition that can disrupt sleep
* women only: irregular menstrual periods or pregnancy
* use of medications/compounds that can disrupt sleep

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Plamen D Penev, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Investigator left academia and is unavailable; participation in cross-over sequences was not unblinded, therefore participants are presented in one Arm throughout Results.
Period: Overall Study
Arm/Group | Eszopiclone or Placebo
Started | 20
Completed | 16
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eszopiclone or Placebo
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Plasma Glucose Level at the 120-minute Time Point of a 75g Oral Glucose Tolerance Test
Time Frame: at the end of each treatment
Population: Investigator left university without analyzing data and no information is available on unblinding.
Arm/Group | Eszopiclone or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Eszopiclone or Placebo
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eszopiclone or Placebo (N=20)
Furuncle (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes